CLINICAL TRIAL: NCT03731637
Title: A Prospective Study to Establish a New Onset Hyperglycemia and Diabetes (NOD) Cohort
Brief Title: A Study to Establish a New Onset Hyperglycemia and Diabetes Cohort
Acronym: NOD
Status: Terminated | Type: Observational
Why Stopped: Low recruitment rate and low event rate (pancreatic cancer).
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Principal Investigator, Ziding Feng, Professor, Fred Hutchinson Cancer Center
Other Study IDs: 17-011305; U01DK108328 (NIH); A211701 (Other: CTEP Identifier); NCI-2018-01307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1001811 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Type2 Diabetes; Diabetes Mellitus
Keywords: New Onset Diabetes; Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research Blood Collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- New-onset diabetes: Subjects with biochemically-defined new-onset diabetes

SUMMARY:
Create a large biobank of blood samples and data from subjects with new onset hyperglycemia and diabetes (NOD).

DETAILED DESCRIPTION:
A prospective NOD Cohort of 10,000 eligible, enrolled subjects will be assembled over the next 5 years, with each patient participating for up to 3 years from the date they meet biochemical (glycemic) criteria for diabetes. Sites electronic medical record databases or other avenues for recruitment, such as physician and self referral, will be utilized to identify subjects meeting criteria for NOD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to provide informed consent and sign an informed consent form.
* Subject must sign an authorization for the release of their protected health information.
* Subject must be ≥50 and ≤85 years of age at the time of enrollment.
* Subject must have hyperglycemia and/or diabetes as one of the following within 90 days prior to enrollment:

  * All glycemic parameters must be measured in an outpatient setting

A. (1) Hemoglobin A1c (HbA1c) ≥ 6.5% present, OR

B. Any (2) PDMs present on consecutive or simultaneous testing:

* Fasting Blood Glucose (FBG) ≥126 mg/dl
* Hemoglobin A1c (HbA1c) ≥ 6.5%
* Random Blood Glucose (RBG) ≥200 mg/dl
* 2h Post Glucose (PG) ≥200mg (11.1 mmol/L) during OGTT (oral glucose tolerance test), OR

C. Any (1) PDM present followed by an anti-diabetes medication

* Subject must have >1 glycemic parameter measured in the 18 months prior to the elevated index lab without meeting inclusion criteria A, B, or C.
* Subject must be willing to provide blood samples (fasting) at baseline, 6, 12, and 24 months post-enrollment.
* Subject or authorized representative must be willing to complete a detailed questionnaire.

Exclusion Criteria:

* Subject must not have any past history of hyperglycemia and/or diabetes as defined by inclusion criteria A, B, or C

  * Transient diabetes (e.g. gestational and steroid-induced) is not an exclusion.
* Subject must not be on active treatment for cancer, carry a current diagnosis of any cancer, and/or investigated for suspicion of recurrence of past cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix).

  * Ongoing work up for suspicion of pancreatic cancer is not an exclusion.
* Subject must not have any past history of pancreatic cancer.
* Subject must not be on anti-diabetes medications prior to the elevated index lab.
* Subject must not be on chronic or acute use of steroid medications within 90 days of the elevated index lab.

  * Allowed: Nasal, topical steroids, oral budesonide, ophthalmic
* Subject must not have had a recent (within 1 week of the elevated index lab) intra-articular steroid injection.
* In the physician's and/or investigator's judgement, subject does not have any co-morbidities that limit the subject's participation in the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who newly meet criteria for diabetes
Sampling Method: Probability Sample
Enrollment: 2269 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pancreatic ductal adenocarcinoma in new-onset hyperglycemia and diabetes | 3 years
  Enrolled subjects will be followed for three years to determine the 1-year, 2-year, 3-year incidence rates of PDAC in new-onset hyperglycemia and diabetes.
Determine sensitivity and specificity of serum CA 19-9 in pre-symptomatic pancreatic ductal adenocarcinoma in subjects with new-onset hyperglycemia and diabetes | 3 years
  We will retrospectively measure serum CA 19-9 in blood collected at baseline and at each subsequent blood draw to determine its ability to predict pancreatic cancer in presymptomatic subjects. We will also collect blood for future biomarker testing.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Chari, MD, Study Chair — M.D. Anderson Cancer Center; Anirban Maitra, MBBS, Study Chair — M.D. Anderson Cancer Center; Bechien Wu, MD, Study Chair — Kaiser Permanente Southern Califorina
Locations (18):
- United States (18):
  - Kaiser Permanente Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Greater Los Angeles Veterans Affairs Medical Center, Los Angeles, California
  - Kaiser Permanente Northern California, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Advent Health Translational Research Institute, Orlando, Florida
  - Carle Foundation Hospital, Urbana, Illinois
  - Univeristy Hospital, Indiana University Health, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Trinity Health Ann Arbor Hospital, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Marshfield Clinic Health System, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chari ST, Leibson CL, Rabe KG, Ransom J, de Andrade M, Petersen GM. Probability of pancreatic cancer following diabetes: a population-based study. Gastroenterology. 2005 Aug;129(2):504-11. doi: 10.1016/j.gastro.2005.05.007. PMID 16083707
- [Background] Sharma A, Smyrk TC, Levy MJ, Topazian MA, Chari ST. Fasting Blood Glucose Levels Provide Estimate of Duration and Progression of Pancreatic Cancer Before Diagnosis. Gastroenterology. 2018 Aug;155(2):490-500.e2. doi: 10.1053/j.gastro.2018.04.025. Epub 2018 Apr 30. PMID 29723506
- [Background] Setiawan VW, Stram DO, Porcel J, Chari ST, Maskarinec G, Le Marchand L, Wilkens LR, Haiman CA, Pandol SJ, Monroe KR. Pancreatic Cancer Following Incident Diabetes in African Americans and Latinos: The Multiethnic Cohort. J Natl Cancer Inst. 2019 Jan 1;111(1):27-33. doi: 10.1093/jnci/djy090. PMID 29917105
- [Derived] Chari ST, Maitra A, Matrisian LM, Shrader EE, Wu BU, Kambadakone A, Zhao YQ, Kenner B, Rinaudo JAS, Srivastava S, Huang Y, Feng Z; Early Detection Initiative Consortium. Early Detection Initiative: A randomized controlled trial of algorithm-based screening in patients with new onset hyperglycemia and diabetes for early detection of pancreatic ductal adenocarcinoma. Contemp Clin Trials. 2022 Feb;113:106659. doi: 10.1016/j.cct.2021.106659. Epub 2021 Dec 23. PMID 34954100
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials